CLINICAL TRIAL: NCT01789762
Title: Evaluation of the Efficacy of Platelets Treated With Pathogen Reduction Process
Acronym: EFFIPAP
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Etablissement Français du Sang (Other)
Collaborators: University Hospital, Grenoble (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 2012-P001
Record Dates: First submitted 2013-02-08; First posted 2013-02-12 (Estimated); Last update posted 2019-04-29 (Actual); Status verified 2016-08

CONDITIONS: Aplasia With Expected Thrombocytopenia
Keywords: Platelet transfusions; Pathogen reduction; Haemorrhagic episodes

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Historical control arm (Active Comparator): Patients transfused with platelet concentrates re-suspended in autologous plasma
  Interventions: Biological: Autologous plasma
- Control arm (Active Comparator): Patients transfused with platelets prepared in additive solution
  Interventions: Biological: Additive solution
- Experimental arm (Experimental): Patients transfused with platelets treated by pathogen reduction process
  Interventions: Biological: Pathogen reduction process

INTERVENTIONS:
Biological: Autologous plasma — Transfusions of platelet concentrates re-suspended in autologous plasma
  Arms: Historical control arm
Biological: Additive solution — Transfusions of platelets prepared in additive solution (Intersol)
  Arms: Control arm
Biological: Pathogen reduction process — Patients transfused with platelets treated by pathogen reduction process
  Arms: Experimental arm

SUMMARY:
This study is a multicentre, double-blind, randomized therapeutic trial.

The primary objective of this study is to evaluate non-inferiority with regard to prevention and control of haemorrhage:

* of platelet concentrates treated by pathogen reduction(Intercept amotosalen and UVA procedure)
* compared with the usual platelet concentrates (in additive solution intersol), reference arm, and
* compared with platelet concentrates re-suspended in autologous plasma (historic arm) These three products are available and authorised by ANSM (formerly AFSSAPS).

The secondary objectives is to evaluate the transfusion needs, transfusion outcomes and safety and the decreased frequency of grade 2 or higher side effects related to transfusion allergy to platelets.

DETAILED DESCRIPTION:
There is an unresolved difficulty in the evaluation of haemorrhagic symptoms in thrombocytopenia due to the very nature of the scale, which is the international standard at this time (WHO scale). This scale is based on the level of blood loss and is applicable to any haemostasis disorder. We will keep it as the standard but have decided to be particularly rigorous in the data collection and will perform daily haemorrhagic assessment.

Several sequences of missing data can be imputed for one patient. Each sequence of missing data will be replaced if and only if the number of consecutive days missing does not exceed 15%* of the total length of the patient's stay. If one sequence of missing data is longer than the 15%, no replacement will be done for the patient. (Example: If the total stay is 30 days, the maximal length of a missing data sequence accepted is 4 days). The following strategies will be used to replace missing data:

• The first observation is missing: Next observation carried backwards (NOCB) assigns the next known score after the missing value to the missing one.

• The last observation is missing: Last observation carried forward (LOCF) assigns the last known score before the missing value to the missing one. (Suppose that the situation is stable whilst the patient is leaving the hospital.)

• Sequence of one or several missing data with non-missing data before and after the sequence: Last and Next1 assigns the average of the person's last known and next known observation to the missing value. The score is rounded down to the nearest whole number if needed. (Ex mean (1+2) =1)

* 15% rounded up to nearest whole number.

1 : Engels, J.M. 2003. Imputation of Missing Longitudinal Data : a Comparison of Methods. Journal of Clinical Epidemiology 56 (2003) 968-976

Following a quality analysis of EFFIPAP study's recruitment, it was decided by the sponsor to increase the number of patients. Approximatively thirty additional patients will be included in order to replace non analyzable patients for the following reasons : wrongly included, non-transfused patients, consent withdrawal. Those 30 additional patients will allow us to reach our initial target of 810 analyzable patients in order to respond to the main objective of the study

ELIGIBILITY:
Inclusion Criteria:

* Patients aged 18 years or older
* Patient hospitalised for bone marrow aplasia, with expected stay of over 10 days and in principle requiring platelet transfusion support (at least twice).
* Signed informed consent
* Patients with DIC can be included; they will undergo a separate analysis.
* A negative pregnancy test is necessary before inclusion in all women of childbearing age

Exclusion Criteria:

* Patient included in this trial previously during a prior aplasia episode.
* Patient requiring curative anticoagulant treatment at the time of inclusion (vitamin K antagonists, heparin (LMWH and NFH), anti-IIa and Xa at curative doses for treatment or prophylaxis of arterial or venous thromboembolic disease (TED) or as part of the treatment for cardiac valvulopathy and complications of atrial fibrillation).
* Thrombocytopenia due to increased destruction
* Patient requires washed platelet concentrates (i.e., with residual plasma less than that remaining during the addition of an additive solution) due to previous intolerance to platelets (cf IgA deficiency, history of major allergic reaction)
* Patient requiring products "CMV negative " (previously included in a protocol transfusion CMV negative)
* Patients with platelet transfusion refractoriness during a previous period of cytopenia, including patient with platelet refractoriness related to an anti-HLA alloimmunization (thus, patient already known as requiring compatible platelets HLA)
* Patient who requires compatible HLA platelets due to a refractory state relative to anti-HLA alloimmunization
* Patient presenting a platelet transfusion refractoriness at the time of previous aplasia.
* Protected adults and persons deprived of liberty

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 842 (Actual)
Dates: Start 2013-05; Primary Completion 2016-01 (Actual); Study Completion 2016-01 (Actual)

PRIMARY OUTCOMES:
Incidence of grade 2 or higher (WHO) haemorrhagic episodes | During 1 month

SECONDARY OUTCOMES:
Frequency incidence of haemorrhagic episodes (grade 1 and higher) | During 1 month
Number of serious grade 3-4 haemorrhagic episodes | During 1 month
Number of minor grade 1 haemorrhagic episodes | During 1 month
Transfusion outcome in platelets (CCI) at 24 hours | During 1 month
Number of transfusions of platelet concentrates and red blood cells | During 1 month
Transfusion intervals | During 1 month
Safety (transfusion side effects) grade 2 or higher | During 1 month
Occurrence of anti-platelet antibodies (Anti-HLA, anti-HPA) | During 1 month
Occurrence of platelet transfusions refractiveness | During 1 month
Validation of a new haemorrhagic evaluation: EFS scale | During 1 month
Variation in hematocrit and hemoglobin levels | During 1 month

CONTACTS AND LOCATIONS:
Locations (12):
- France (12):
  - CHU de Besancon, Besançon
  - CHU de Brest, Brest
  - CHU de Clermont Ferrand, Clermont-Ferrand
  - CHU Henri Mondor - APHP, Créteil
  - CHU de Dijon, Dijon
  - CHU de Grenoble, Grenoble
  - Hopital Huriez - CHRU Lille, Lille
  - Institut Paoli Calmette, Marseille
  - Hopital Saint Antoine, Paris
  - Hospices Civils de Lyon - Lyon Sud, Pierre-Bénite
  - CHU de Rennes, Rennes
  - Institut de Cancérologie de la Loire, Saint-Priest-en-Jarez

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Garban F, Guyard A, Labussiere H, Bulabois CE, Marchand T, Mounier C, Caillot D, Bay JO, Coiteux V, Schmidt-Tanguy A, Le Niger C, Robin C, Ladaique P, Lapusan S, Deconinck E, Rolland C, Foote AM, Francois A, Jacquot C, Tardivel R, Tiberghien P, Bosson JL; Evaluation of the Efficacy of Platelets Treated With Pathogen Reduction Process (EFFIPAP) Study Group. Comparison of the Hemostatic Efficacy of Pathogen-Reduced Platelets vs Untreated Platelets in Patients With Thrombocytopenia and Malignant Hematologic Diseases: A Randomized Clinical Trial. JAMA Oncol. 2018 Apr 1;4(4):468-475. doi: 10.1001/jamaoncol.2017.5123. PMID 29392283